CLINICAL TRIAL: NCT02894671
Title: Ischemia Modified Albumin (IMA) Expression in the Male and Female Population
Acronym: IMAandGENDER
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Giovanni Bracci, MD, Istituto Ortopedico Rizzoli
Other Study IDs: 83/14
Record Dates: First submitted 2016-02-12; First posted 2016-09-09 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Group Identification
MeSH Terms: conditions — Social Identification

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum vials
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- male under 45y: blood exams performed on males under 45years (in a range of 20-90 years) not wearing articular devices, without fractures, and without these diseases: oncologic, hemochromatosis, hepatic, thalassaemia, diabetes, anemia (Hb<9)
  Interventions: Other: blood exams
- male over 45y: blood exams performed on males over 45years (in a range of 20-90 years) not wearing articular devices, without fractures, and without these diseases: oncologic, hemochromatosis, hepatic, thalassaemia, diabetes, anemia (Hb<9)
  Interventions: Other: blood exams
- fertile female: blood exams performed on fertile females (in a range of 20-90 years) not wearing articular devices, no pregnant, without fractures, and without these diseases: oncologic, hemochromatosis, hepatic, thalassaemia, diabetes, anemia (Hb<9)
  Interventions: Other: blood exams
- infertile female: blood exams performed on infertile females (in a range of 20-90 years) not wearing articular devices, no pregnant, without fractures, and without these diseases: oncologic, hemochromatosis, hepatic, thalassaemia, diabetes, anemia (Hb<9)
  Interventions: Other: blood exams

INTERVENTIONS:
Other: blood exams — in serum will be analyzed the level of IMA, iron, transferrin, ferritin, total albumin

SUMMARY:
The study has as general objective to analyze in the adult population, (male and female) the presence of a very common protein, in its normal form and modified, isolated from the blood of patients and called albumin. The opportunity to observe the distribution of this protein in the population, provides the basis to be able to perform this type of assay also in the population of patients with pathologies, in the near future, with the aim of increasing knowledge on the subjective tolerability to orthopedic implants.

DETAILED DESCRIPTION:
100 patients, waiting for elective surgical intervention (such as hip replacement or primary knee ligament reconstruction, arthroscopy), distributed evenly by gender and age (50 men, 50 women including 25 postmenopausal and 25 in bearing age) and afferent to the Department of Surgery Prosthetic hip and knee of our Institute, will be enrolled. At execution time of blood sampling routine, a further specimen of whole blood (7 ml) will be added which will be sent to the Medical technology laboratory for IMA dosage. In addition, total albumin, ferritin, transferrin and serum iron will be analyzed from clinical pathological laboratory. The investigators will be able to analyze the IMA and normalized IMA distributions with respect to gender factor and correlation with the three listed blood tests (ferritin, transferrin and serum iron).

ELIGIBILITY:
* Inclusion Criteria:
* caucasic
* signed informative consensus
* Exclusion Criteria:
* patients wearing articular devices
* pregnant (for female)
* fractured patients
* patients with oncologic diseases, hemochromatosis, hepatic diseases, thalassaemia, diabetes, anemia (Hb<9)

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 25 males under 45y, 25 males over 45y, 25 fertile females and 25 infertile females
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
IMA dosage | one year
  Dosage of IMA (mg/ml), with ELISA assay for each patient

SECONDARY OUTCOMES:
iron, transferrin dosages | one year
  Dosage of iron and transferrin (mg/ml) values in patients blood
Ferritin dosages | one year
  Dosage of ferritin (ng/ml) values in patients blood

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Bracci, MD, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli - Laboratorio Tecnologia Medica, Bologna, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Govender R, De Greef J, Delport R, Becker PJ, Vermaak WJ. Biological variation of ischaemia-modified albumin in healthy subjects. Cardiovasc J Afr. 2008 May-Jun;19(3):141-4. PMID 18568173
- [Background] Catalani S, Leone R, Rizzetti MC, Padovani A, Apostoli P. The role of albumin in human toxicology of cobalt: contribution from a clinical case. ISRN Hematol. 2011;2011:690620. doi: 10.5402/2011/690620. Epub 2010 Oct 31. PMID 22084701
- [Background] Bar-Or D, Rael LT, Lau EP, Rao NK, Thomas GW, Winkler JV, Yukl RL, Kingston RG, Curtis CG. An analog of the human albumin N-terminus (Asp-Ala-His-Lys) prevents formation of copper-induced reactive oxygen species. Biochem Biophys Res Commun. 2001 Jun 15;284(3):856-62. doi: 10.1006/bbrc.2001.5042. PMID 11396981